CLINICAL TRIAL: NCT03707951
Title: A Proof-of-Concept Trial of N-Acetylcysteine for Adolescent Alcohol Use Disorder
Brief Title: N-Acetylcysteine for Adolescent Alcohol Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Kevin Gray, Professor of Psychiatry and Behvavioral Sciences, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO#00080921
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Alcohol Use Disorder
Keywords: alcohol; youth; adolescent; pharmacotherapy; medication; N-acetylcysteine
MeSH Terms: conditions — Alcoholism | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: 1:1 parallel group allocation randomized placebo controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind placebo-controlled pharmacotherapy trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- N-acetylcysteine (Experimental): N-acetylcysteine 1200 mg twice daily for 8 weeks; administered orally
  Interventions: Drug: N-acetylcysteine
- Placebo (Placebo Comparator): Placebo (matched in appearance to N-acetylcysteine to preserve double-blind) twice daily for 8 weeks; administered orally
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: N-acetylcysteine — N-acetylcysteine 1200 mg twice daily for 8 weeks (administered orally)
  Arms: N-acetylcysteine
Drug: Placebo oral capsule — Placebo (matched in appearance to N-acetylcysteine to preserve double-blind) twice daily for 12 weeks (administered orally)
  Arms: Placebo

SUMMARY:
This is a 8-week randomized, placebo-controlled trial testing the effects of N-acetylcysteine (NAC), on a platform of weekly evidence-based brief alcohol intervention for 120 adolescents with alcohol use disorder (AUD). The primary efficacy endpoint is reduction in alcohol use (total standard drinks), compared between NAC and placebo groups.

DETAILED DESCRIPTION:
Adolescence is a critical developmental stage involving marked elevation in alcohol initiation, progression to AUD, and development of significant, lasting adverse outcomes from use. Effective treatments must be developed for AUD in this especially vulnerable age range. The identification of a well-tolerated, effective pharmacological treatment would represent a significant advance and could yield tremendous public health impact. The proposed trial will provide critical data to evaluate NAC as a highly promising pharmacotherapy for adolescent AUD, and regardless of NAC versus placebo outcomes will provide key methodological guidance for future randomized controlled trials of pharmacotherapies for adolescent AUD. Randomized participants will be provided and instructed to take their assigned medication at 1200 mg twice daily, in approximately twelve-hour intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 13-25
2. Must be able to understand the study and provide written informed consent (for participants under 18 years old, a parent/legal guardian must be able to provide consent and the participant must be able to provide assent).
3. Current moderate to heavy drinker by established adolescent criteria
4. Meet criteria for alcohol use disorder
5. Females must agree to use appropriate birth control methods during study participation: oral contraceptives, contraceptive patch, barrier (diaphragm or condom), levonorgestrel implant, medroxyprogesterone acetate, complete abstinence from sexual intercourse, or hormonal contraceptive vaginal ring

Exclusion Criteria:

1. Score >10 on the Clinical Institute Withdrawal Assessment for Alcohol
2. Allergy or intolerance to N-acetylcysteine
3. Females who are pregnant, contemplating pregnancy or lactating over the next 6 months
4. Current use of N-acetylcysteine or any supplement containing N-acetylcysteine (must agree not to take any such supplement throughout study participation)
5. Current enrollment in treatment for alcohol use disorder or expectation of other treatment during protocol participation
6. Any other medical or psychiatric condition or other significant concern that in the Investigator's opinion would impact participant safety or compliance with study instructions, or potentially cofound the interpretation of findings

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 126 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Gray, MD, Principal Investigator — Professor of Psychiatry and Behavioral Sciences
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Squeglia LM, Tomko RL, Baker NL, Kirkland AE, McClure EA, Gray KM. A Randomized Controlled Trial of N-acetylcysteine for Adolescent and Young Adult Alcohol Use Disorder. J Am Acad Child Adolesc Psychiatry. 2025 Sep 26:S0890-8567(25)02088-X. doi: 10.1016/j.jaac.2025.09.025. Online ahead of print. PMID 41016625

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | N-acetylcysteine | Placebo
Started | 65 | 61
Completed Active Treatment | 53 | 52
Completed | 51 | 38
Not Completed | 14 | 23
Not completed — Lost to Follow-up | 8 | 17
Not completed — Withdrawal by Subject | 6 | 6

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | N-acetylcysteine | Placebo | Total
Number analyzed (Participants) | 65 | 61 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.1 (2.3) | 20.9 (2.4) | 21.0 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 37 | 78
  Male | 24 | 24 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 62 | 55 | 117
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 58 | 53 | 111
  More than one race | 3 | 5 | 8
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 65 | 61 | 126

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Use During the Final 4 Weeks of Treatment (Weeks 5 - 8)
Description: Alcohol use (total standard drinks) during the final four weeks of treatment (Weeks 5-8), compared between NAC and placebo groups.
Time Frame: Final 4 weeks of treatment
Population: Randomized participants
Measure: Mean (Standard Deviation); unit: Standard drinks
Arm/Group | N-acetylcysteine | Placebo
Number analyzed (Participants) | 65 | 61
Standard drinks | 37.9 (28.3) | 42.6 (43.1)

ADVERSE EVENTS:
Time Frame: 6 months (from randomization to final post-treatment follow-up visit)
Description: Adverse events were assessed and documented by the study medical clinician and entered using MedDRA terminology.
Arm/Group | N-acetylcysteine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/61
Other Adverse Events (participants affected / at risk) | 48/65 | 41/61
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-acetylcysteine (N=65) | Placebo (N=61)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Otitis media (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 3 (3)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (2)
Decreased appetite (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 9 (15) | 1 (1)
Dyspepsia (worsening) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5 (6) | 2 (2)
Nausea (Gastrointestinal disorders) | 12 (14) | 12 (16)
Regurgitation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary gland calculus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomachache (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (4)
Dysguesia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (4) | 2 (2)
Malaise (General disorders) | 0 (0) | 1 (1)
Pain in jaw (General disorders) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 3 (3) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Influenza-like illness (Infections and infestations) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (3) | 1 (1)
Pharyngitis, streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Sinus headache (Infections and infestations) | 1 (1) | 0 (0)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 2 (2)
Vaginal infection (Infections and infestations) | 3 (3) | 1 (1)
Viral upper respiratory infection (Infections and infestations) | 12 (15) | 8 (9)
Accidental exposure to product (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Weight increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Body aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Restless leg syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Concussion (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 10 (12) | 11 (14)
Hypothesia (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Paresthesias (Nervous system disorders) | 3 (3) | 1 (1)
Sleep paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Vivid dreams (Nervous system disorders) | 0 (0) | 2 (2)
Menstruation delayed (General disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Anxiety (worsening) (Psychiatric disorders) | 3 (3) | 2 (2)
Attention-Deficit/Hyperactivity Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (6) | 7 (8)
Mood swings (Psychiatric disorders) | 0 (0) | 1 (1)
Post-operative pain (General disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysmenorrhea (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Irregular menses (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Mastalgia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Oopharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Seasonal rhinitis (worsening) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus headache (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sunburn (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Post-procedural complication (Surgical and medical procedures) | 1 (1) | 0 (0)
Post-operative pain (Surgical and medical procedures) | 1 (1) | 0 (0)
Tonsillectomy/uvulectomy (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-11): https://cdn.clinicaltrials.gov/large-docs/51/NCT03707951/Prot_SAP_001.pdf